CLINICAL TRIAL: NCT00377767
Title: Improving Primary Care to Prevent Childhood Obesity
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: R01HD050966 (NIH)
Record Dates: First submitted 2006-09-15; First posted 2006-09-18 (Estimated); Last update posted 2006-09-18 (Estimated); Status verified 2006-09

CONDITIONS: Overweight in Preschool Age Children; Risk of Overweight in Preschool Age Children
Keywords: Chronic Care Model; Obesity; Overweight; Children; Body Mass Index; Primary Care
MeSH Terms: conditions — Obesity; Overweight

INTERVENTIONS:
Behavioral: To change structure and roles of primary care teams to optimize prevention of obesity

SUMMARY:
To determine the extent to which a clinical intervention based on the Chronic Care Model (CCM), compared with the usual care control condition, results in a smaller age-associated increase in body mass index (BMI) over a 1 year intervention (primary outcome) and a 1 1/2-year follow-up period.

DETAILED DESCRIPTION:
Overweight in the preschool age group is prevalent, increasing, and of consequence. During the last 30 years in the U.S., the prevalence of overweight among youth has dramatically increased. Overweight in young children is associated with later overweight, with childhood conditions such as hyperlipidemia, hypertension, and type II diabetes, and with higher morbidity and mortality in adulthood.

Along with the long-term risks associated with overweight in the preschool age group, there come unique opportunities to intervene and alter the subsequent course of health and disease for these individuals. These regular visits allow both detection of elevated BMI levels and opportunities for intervention.

The overall goal of this research is to assess a comprehensive, innovative, primary care practice change intervention to prevent obesity among children age 2 through 5 years at elevated risk of obesity. To achieve this goal, we will conduct a cluster-randomized controlled trial in 10 pediatric practices of Harvard Vanguard Medical Associates, a large multi-site group practice in eastern Massachusetts with a track record of research collaboration.

We will randomize five health centers to the intervention condition, and five health centers to the control (usual care) condition. The intervention will consist of state-of-the-science approaches to changing dietary, activity, and inactivity behaviors among the children.

The intervention period will be 1 year, followed by a 1 1/2 year maintenance follow-up period. Frequency of visits will be every 6 weeks for the first 6 months, and every 6 months after that. Participating families will complete a telephone-administered interview at baseline and all follow-up timepoints. There will be 3 types of measurements: 1) measurements made by the clinical staff that will also be used for outcomes in the research study (only height and weight); 2) measurements made by clinicians for feedback during counseling sessions, which will not be used for study outcomes; and 3) measurements made by the research staff for study outcomes and processes.

ELIGIBILITY:
Inclusion Criteria:

* Age 2.0 through 5.9 years receiving primary care in a multi-site group practice
* BMI > 95th percentile for age and sex, or 85th - 95th percentile if at least one parent is overweight

Exclusion Criteria:

* Child currently enrolled in a formal weight management program
* Child is in foster care
* Chronic conditions that may limit our ability to measure height and weight or that may interfere with their growth, physical activity, or dietary recommendations

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500
Dates: Start 2006-09; Study Completion 2009-09

PRIMARY OUTCOMES:
Body mass index (BMI) at 1 year.

SECONDARY OUTCOMES:
Television viewing behaviors at 1 year post intervention.
Sugar-sweetened beverages intake at 1 year post intervention.
Fast food intake at 1 year post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Gillman, MD, Principal Investigator — Department of Ambulatory Care and Prevention/Harvard Pilgrim Health Care/ Harvard Medical School
Locations (1):
- Harvard Vanguard Medical Associates, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Wright DR, Taveras EM, Gillman MW, Horan CM, Hohman KH, Gortmaker SL, Prosser LA. The cost of a primary care-based childhood obesity prevention intervention. BMC Health Serv Res. 2014 Jan 29;14:44. doi: 10.1186/1472-6963-14-44. PMID 24472122
- [Derived] Hohman KH, Price SN, Sonneville K, Rifas-Shiman SL, Gortmaker SL, Gillman MW, Taveras EM. Can the Internet be used to reach parents for family-based childhood obesity interventions? Clin Pediatr (Phila). 2012 Apr;51(4):314-20. doi: 10.1177/0009922811423310. Epub 2011 Oct 12. PMID 21997144
- [Derived] Taveras EM, Gortmaker SL, Hohman KH, Horan CM, Kleinman KP, Mitchell K, Price S, Prosser LA, Rifas-Shiman SL, Gillman MW. Randomized controlled trial to improve primary care to prevent and manage childhood obesity: the High Five for Kids study. Arch Pediatr Adolesc Med. 2011 Aug;165(8):714-22. doi: 10.1001/archpediatrics.2011.44. Epub 2011 Apr 4. PMID 21464376
- [Derived] Taveras EM, Hohman KH, Price SN, Rifas-Shiman SL, Mitchell K, Gortmaker SL, Gillman MW. Correlates of participation in a pediatric primary care-based obesity prevention intervention. Obesity (Silver Spring). 2011 Feb;19(2):449-52. doi: 10.1038/oby.2010.207. Epub 2010 Sep 16. PMID 20847735